CLINICAL TRIAL: NCT05497557
Title: An Open-label Study to Evaluate the Impact of Omeprazole, A Proton Pump Inhibitor, on the Pharmacokinetics of Sotorasib Co-administered With an Acidic Beverage in Healthy Volunteers
Brief Title: A Study to Evaluate the Impact of Omeprazole on the Pharmacokinetics of Sotorasib Co-administered With an Acidic Beverage in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20220024
Record Dates: First submitted 2022-08-03; First posted 2022-08-11 (Actual); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Sotorasib; AMG 510; Omeprazole
MeSH Terms: interventions — Omeprazole; sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omeprazole + Sotorasib (Experimental)
  Interventions: Drug: Omeprazole; Drug: Sotorasib

INTERVENTIONS:
Drug: Omeprazole — Omeprazole will be administered as an oral capsule.
Drug: Sotorasib — Sotorasib will be administered as an oral tablet.
  Other Names: AMG 510

SUMMARY:
The primary objective of the study is to evaluate the effects of omeprazole (a proton-pump inhibitor) and an acidic beverage (Coca-Cola) on sotorasib pharmacokinetics (PK) when administered orally in healthy volunteers.

ELIGIBILITY:
Inclusion:

* Healthy male participants or female participants, between 18 and 60 years of age (inclusive), at the time of Screening.
* Body mass index, between 18 and 30 kg/m^2 (inclusive), at the time of Screening.
* Females of nonchildbearing potential.

Exclusion:

* Inability to swallow oral medication or history of malabsorption syndrome.
* History of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
* Poor peripheral venous access.
* History or evidence, at Screening or Check in, of clinically significant disorder, condition, or disease, including history of myolysis, not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Labcorp Clinical Research Unit Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 16 participants were enrolled at 1 center in the United States.
Pre-assignment Details: Participants were screened to assess their eligibility to enter the study within 28 days prior to the first dose administration.
Groups:
- Sotorasib Alone: On Day 1, participants received 960 mg sotorasib (8 x 120 mg tablets) administered orally with 240 mL of water after an overnight fast of at least 10 hours.
- Omeprazole Alone: On Days 4 to 8, participants received 40 mg omeprazole (delayed release capsule) administered orally with 240 mL of water once daily (QD) after an overnight fast of at least 10 hours.
- Omeprazole Co-administered With Sotorasib: On Day 9, participants received 40 mg omeprazole (delayed release capsule) followed by 960 mg sotorasib (8 x 120 mg tablets) administered orally within 5 minutes with 240 mL of an acidic beverage after an overnight fast of at least 10 hours.
Period: Period 1: Sotorasib Alone
Arm/Group | Sotorasib Alone | Omeprazole Alone | Omeprazole Co-administered With Sotorasib
Started | 16 | 0 | 0
Completed (Participants who completed Period 1, in which they received sotorasib alone on Day 1. All completed participants continued onto Period 2.) | 16 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Period 2: Omeprazole Alone
Arm/Group | Sotorasib Alone | Omeprazole Alone | Omeprazole Co-administered With Sotorasib
Started | 0 | 16 | 0
Completed (Participants who completed Period 2, in which they received omeprazole alone on Days 4 to 8. All completed participants continued onto Period 3.) | 0 | 14 | 0
Not Completed | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0
Period: Period 3: Omeprazole With Sotorasib
Arm/Group | Sotorasib Alone | Omeprazole Alone | Omeprazole Co-administered With Sotorasib
Started | 0 | 0 | 14
Completed (Participants who completed Period 3, in which they received omeprazole co-administered with sotorasib on Day 9.) | 0 | 0 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented in the All Subjects Population, which included all participants who signed the informed consent form and had any study assessment recorded in the database per the protocol.
Groups:
- Sotorasib and Omeprazole: All Participants: On Day 1, participants received 960 mg sotorasib (8 x 120 mg tablets) administered orally with 240 mL of water after an overnight fast of at least 10 hours. On Days 4 to 8, participants received 40 mg omeprazole (delayed release capsule) administered orally with 240 mL of water QD after an overnight fast of at least 10 hours. On Day 9, participants received 40 mg omeprazole (delayed release capsule) followed by 960 mg sotorasib (8 x 120 mg tablets) administered orally within 5 minutes with 240 mL of an acidic beverage after an overnight fast of at least 10 hours.
Arm/Group | Sotorasib and Omeprazole: All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Sotorasib
Time Frame: Predose (Hour 0), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, and 48 hours postdose following administration of sotorasib on Days 1 and 9
Population: Measured in the Pharmacokinetic Population for the primary endpoint analyses, which included all participants who received both sotorasib, and sotorasib in combination with omeprazole and an acidic beverage, and had evaluable pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Sotorasib Alone | Omeprazole Co-administered With Sotorasib
Number analyzed (Participants) | 16 | 14
ng/mL | 7160 (22.9) | 4850 (65.6)
Statistical Analysis 1: Comparison: Sotorasib Alone vs Omeprazole Co-administered With Sotorasib; Ratios of geometric least squares means, and corresponding confidence intervals were obtained by taking the exponential of the least square means (LSMs), differences in LSMs, and corresponding confidence intervals on the natural log (ln) scale; Test type: Other — Drug-drug Interaction Assessment; Ratio of geometric least squares mean = 0.677, 90% CI 2-sided [0.547 to 0.839]

2. Primary Outcome: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUCinf) of Sotorasib
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sotorasib Alone | Omeprazole Co-administered With Sotorasib
Number analyzed (Participants) | 16 | 14
h*ng/mL | 30200 (33.3) | 23500 (60.4)
Statistical Analysis 1: Comparison: Sotorasib Alone vs Omeprazole Co-administered With Sotorasib; [analysis description as in outcome 1, analysis 1]; Test type: Other — Drug-drug Interaction Assessment; Ratio of geometric least squares mean = 0.771, 90% CI 2-sided [0.628 to 0.948]

3. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-tlast) of Sotorasib
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Sotorasib Alone | Omeprazole Co-administered With Sotorasib
Number analyzed (Participants) | 16 | 14
h*ng/mL | 30000 (33.3) | 23200 (62.2)
Statistical Analysis 1: Comparison: Sotorasib Alone vs Omeprazole Co-administered With Sotorasib; [analysis description as in outcome 1, analysis 1]; Test type: Other — Drug-drug Interaction Assessment; Ratio of geometric least squares mean = 0.766, 90% CI 2-sided [0.619 to 0.948]

4. Secondary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: An adverse event is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. A TEAE was defined as an adverse event that starts during or after the first dose, or starts prior to the first dose and increases in severity after the first dose. Any clinically significant changes in clinical laboratory tests, 12-lead electrocardiograms and vital signs were recorded as an adverse event.
Time Frame: Day 1 to Day 11
Population: Measured in the Safety Population, which included all participants who received at least 1 dose of study treatment and had at least 1 post-dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sotorasib Alone | Omeprazole Alone | Omeprazole Co-administered With Sotorasib
Number analyzed (Participants) | 16 | 16 | 14
Participants | 0 | 2 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 11
Description: All-cause mortality, serious and other adverse events were measured in the Safety Population, which included all participants who received at least 1 dose of study treatment and had at least 1 post-dose safety assessment.
Arm/Group | Sotorasib Alone | Omeprazole Alone | Omeprazole Co-administered With Sotorasib
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 2/16 | 0/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sotorasib Alone (N=16) | Omeprazole Alone (N=16) | Omeprazole Co-administered With Sotorasib (N=14)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT05497557/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/57/NCT05497557/SAP_001.pdf